CLINICAL TRIAL: NCT01713101
Title: Early Administration of Intravenous Tranexamic Acid for Upper Gastrointestinal Bleeding Prior to Endoscopy
Brief Title: Tranexamic Acid for Upper Gastrointestinal Bleeding
Acronym: TAUGIB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1207-163-002
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Acute Upper Gastrointestinal Hemorrhage
Keywords: Gastrointestinal Hemorrhage; Peptic Ulcer Hemorrhage; Hematemesis; Melena; Tranexamic acid
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Peptic Ulcer Hemorrhage; Hematemesis; Melena

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Early intravenous tranexamic acid administration (Experimental): Early intraveous administration of tranexamic acid
  (1g IV bolus over 10 minutes followed by 1g slow infusion over 8 hours
  Interventions: Drug: Early intravenous tranexamic acid administration
- Placebo group (Placebo Comparator): Normal saline (placebo) administration instead of tranexamic acid solution
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Early intravenous tranexamic acid administration — Initial history taking and physical examination --> enrollment --> 1g bolus over 10 minutes followed slow infusion over 8 hours.
  Other Names: tranexamic acid administration; transamine administration; antifibrinolytics administration
  Arms: Early intravenous tranexamic acid administration
Drug: placebo
  Arms: Placebo group

SUMMARY:
This study is to see whether the early intravenous administration of tranexamic acid improves the outcome of acute upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
Previous studies reported that IV/Oral administration of tranexamic acid improves the outcome upper gastrointestinal bleeding. However, the drug is scarcely used nowadays as those studies are outdated in present clinical field where early endoscopic treatment and PPI administration are considered norm. Although a recent meta-analysis done by Cochrane review group concluded that it improves patient survival, other review articles including "Gut" suggested that a well-designed clinical study is needed for re-evaluation of the efficacy and safety of the drug in current clinical situation. We hypothesized that early administration of the drug will significantly decrease the proportion of patient requiring early endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Chief complaint of hematemesis, melena or hematochezia
2. and objective signs of upper gastrointestinal bleeding

Exclusion Criteria:

1. Pregnant woman, age less than 18
2. Patients whose use of the study drug is contraindicated

   * Increased thromboembolic risk

     * History of thromboembolic disease
     * Alleged inherited thrombophilic disorders
     * Malignancy (except those cured and has not recurred more than two years)
     * Nephrotic syndrome
     * Estrogen use
     * Pregnancy
     * HIT, APA
   * High-risk for cardioembolism

     * Underlying structural heart disease where anticoagulation is indicated
     * Underlying cardiac rhythm disorder where anticoagulation is indicated (e.g. atrial fibrillation/flutter)
   * Possibilities of ongoing DIC

     * Signs and symptoms suggestive of clinically significant infectious disease (e.g. body temperature > 38 degree)
     * Any malignancy except those cured and has not recurred more than two years
   * Patients with history or presence of subarachnoid hemorrhage
   * Acquired color vision impairment, visual loss and retinal venous and arterial occlusions
   * Past history of seizure or organic brain lesion that predispose to seizure disorder
3. Previous history of variceal bleeding
4. Cases where informed consent is unobtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring early endoscopic treatment | Within 24 hours of emergency department visit

SECONDARY OUTCOMES:
Endoscopic signs of bleeding | Within 24 hours of emergency department visit
Length of stay | Within one-month of emergency department visit
Need for urgent endoscopy | Within 24 hours of emergency department visit
Endoscopic procedure time/difficulty | Within 24 hours of emergency department visit
Need for transfusion | Within one-month of emergency department visit
Need for surgery/angiographic intervention | Within one-month of emergency department visit
rate of recurrent bleeding | Within one-month of emergency department visit
death of any cause | Within one-month of emergency department visit
thromboembolic complications | Within one-month of emergency department visit

OTHER OUTCOMES:
Effect modification by hyperfibrinolysis and other coagulation related factors | Variable (within 24-hour and 1-month of emergency department visit)
  Separate analysis looking into the interaction between coagulation function and tranexamic acid effect

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, MD, Study Director — Professor, department of emergency medicine; Sang Hyub Lee, MD, Principal Investigator — Professor, department of internal medicine (gastroenterology); Cheol Min Shin, MD, Principal Investigator — Professor, department of internal medicine (gastroenterology)
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyeongi-do, South Korea